CLINICAL TRIAL: NCT05018585
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Diamyd® to Preserve Endogenous Beta Cell Function in Adolescents and Adults With Recently Diagnosed Type 1 Diabetes, Carrying the Genetic HLA DR3-DQ2 Haplotype
Brief Title: A Phase III Study to Investigate if the Study Drug Diamyd Can Preserve Insulin Production and Improve Glycemic Control in Patients Newly Diagnosed With Type 1 Diabetes
Acronym: DIAGNODE-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Diamyd Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAGNODE-3 (D/P3/21/7); 2024-513304-33-00 (EU CTIS Number)
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus; residual beta cell function; HLA DR3-DQ2; Diabetes Mellitus, Type 1; Autoimmune Diseases; Metabolic Disease; Autoimmune Diabetes; Vitamin D; Immune System Diseases; Insulin Dependent Diabetes; rhGAD65; GAD65; GAD-alum; residual c-peptide; T1D; recent-onset T1D; Type 1 Diabetes; HLA; Diamyd; Diabetes; Newly Diagnosed; New onset; DIAGNODE-3; GAD; Diamyd GAD; Intralymphatic injections; Diabetes immunotherapy; Immunotherapy; Antigen-specific; retogatein
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases; Metabolic Diseases; Immune System Diseases | interventions — Aluminum Hydroxide; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: The study is a 2-arm, randomized, double-blind, placebo-controlled, multicenter, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diamyd (Experimental): Patients will be assigned to receive i) three (3) intralymphatic injections with 4µg Diamyd (rhGAD65) on Days 0, 30, and 60 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day -30 through Day 90)
  Interventions: Biological: Recombinant human glutamic acid decarboxylase (rhGAD65) formulated in Alhydrogel®; Dietary Supplement: Colecalciferol 2000 IU
- Placebo (Placebo Comparator): Patients will be assigned to receive i) three (3) intralymphatic injections of Placebo on Days 0, 30, and 60 and; ii) oral vitamin D 2000 IU/daily for 4 months (from Day -30 through Day 90)
  Interventions: Dietary Supplement: Colecalciferol 2000 IU; Biological: Placebo

INTERVENTIONS:
Biological: Recombinant human glutamic acid decarboxylase (rhGAD65) formulated in Alhydrogel® — Recombinant human glutamic acid decarboxylase (rhGAD65) formulated in Alhydrogel®
  Other Names: Diamyd
  Arms: Diamyd
Dietary Supplement: Colecalciferol 2000 IU — Colecalciferol (vitamin D3) 2000 IU (equivalent to 50 microgram vitamin D3).
  Other Names: Divisun 2000 IU
Biological: Placebo — Placebo for Diamyd, Alhydrogel® only
  Arms: Placebo

SUMMARY:
The objective of DIAGNODE-3 is to evaluate the efficacy and safety of three intranodal injections of 4 μg of Diamyd also known as retogatein compared to placebo, along with oral Vitamin D supplementation, to preserve endogenous beta cell function and influence glycemic parameters in adolescent and adults recently diagnosed with T1D carrying the HLA DR3-DQ2 haplotype.

DETAILED DESCRIPTION:
The study is a 2-arm, randomized, double-blind, placebo-controlled, multicenter, clinical trial. Patients will have the HLA genotyping performed at the first Screening visit (Visit 1A). If the results indicate the patient is carrying the HLA DR3-DQ2 haplotype, then the patient will attend the second Screening visit (Visit 1B) to perform the remaining screening procedures. Eligible patients will receive injections of Diamyd (also known as retogatein) or placebo into an inguinal lymph gland at three occasions, with one month intervals along with oral Vitamin D supplementation. All patients will continue to receive intensive insulin treatment from their personal physicians during the whole study period. Patients will be followed in a blinded manner for a total of 24 months.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in this study only if all of the following criteria apply:

1. Must be capable of providing written, signed, and dated informed consent; and for patients who are minors, age-appropriate assent (performed according to local regulations) and parent/caregiver consent.
2. Males and females aged ≥12 and <29 years old at the time of Screening.
3. Diagnosed with T1D (according to the American Diabetes Association [ADA] classification) ≤6 months at the time of Screening (V1A).
4. Possess the HLA DR3-DQ2 haplotype (all patients will be tested; prior genetic testing results will not be accepted).
5. Fasting C-peptide ≥0.12 nmol/L (≥0.36 ng/mL) on at least one occasion prior to randomization.

   (US ONLY): Fasting C-peptide ≥0.12 - ≤1.5 nmol/L (≥0.36 - ≤4.5 ng/mL) on at least one occasion prior to randomization.
6. Possess detectable circulating GAD65 antibodies (lowest level of detection defined by the method used by the central laboratory).
7. Possess HbA1c levels between 35 to 80 mmol/mol (5.4 to 9.5%) on at least one occasion prior to randomization.
8. Be on a stable basal insulin dose for one month prior to inclusion with limited fluctuation of daily basal insulin requirement based on investigator's assessment. For example, if the average basal insulin dose/kg/24h over a 7-day period compared to the previous 7-day period does not vary more than approximately 20% and/or if the daily basal insulin dose does not vary more than 0.1 U/kg/24h, the dose can be considered stable. Individuals that are diagnosed with T1D according to the ADA classification but are not taking insulin are eligible to participate.
9. i. Females of childbearing potential (FOCBP) must agree to avoid pregnancy and have a negative pregnancy test performed at the required study visits.

FOCBP must agree to use highly effective contraception, during treatment and, until 90 days after the last administration of study medication. Birth control methods, which may be considered as highly effective (e.g., a failure rate of less than 1% per year when used consistently and correctly) include:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * Oral.
  * Intravaginal.
  * Transdermal.
* Progestogen-only hormonal contraception associated with inhibition of ovulation:

  * Oral.
  * Injectable.
  * Implantable.
* Intrauterine device.
* Intrauterine hormone-releasing system.
* Bilateral tubal occlusion.
* Vasectomized partner (vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FOCBP trial patient and that the vasectomized partner has received medical assessment of the surgical success).
* Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient).

  9. ii. Male patients must agree to remain abstinent from heterosexual sex during treatment and for 90 days after treatment or, if sexually active, to use two effective methods of birth control (e.g., male uses a condom and female uses contraception) during and for 90 days after treatment. Acceptable male contraception is as follows:
* Condom (male).
* Abstinence from heterosexual intercourse.
* Vasectomy. The agreement to remain abstinent or use two effective methods of birth control will be clearly defined in the informed consent; the patient or legally authorized representatives (e.g., parents, caregivers, or legal guardians) must sign this specific section.

Exclusion Criteria:

Patients are not eligible to be included in this study if any of the following criteria apply:

1. Participation in any other trial aimed to influence beta cell function from time of diagnosis of T1D.
2. Treatment with any oral or non-insulin injectable anti-diabetic medication or other substance used with the intention to preserve beta cell function (e.g., Verapamil, GABA etc.) within 3 months prior to Randomization.
3. History of maturity-onset diabetes of the young (MODY).
4. Pancreatic surgery, chronic pancreatitis, or other pancreatic disorders that could result in decreased beta cell capacity (e.g., pancreatogenous diabetes).
5. Occurrence of DKA or severe hypoglycemia requiring hospitalization in the period of 90 days prior to Randomization (Visit 2).
6. Signs or symptoms suggesting very poorly controlled diabetes e.g., ongoing weight loss, polyuria or polydipsia.
7. Hematologic condition that would make HbA1c uninterpretable including:

   1. Hemoglobinopathy, with the exception of sickle cell trait or thalassemia minor; or chronic or recurrent hemolysis.
   2. Donation of blood or blood products to a blood bank, blood transfusion or participation in a clinical study requiring withdrawal of >400 mL of blood during the 8 weeks prior to the Screening visit.
   3. Significant iron deficiency anemia.
   4. Heart malformations or vaso-occlusive crisis (VOC) leading to increased turnover of erythrocytes.
8. (US ONLY) Clinically significant abnormal hematology results at the time of Screening, specifically any of the following: white blood cells: < 3.5 x 109/L or >15 x 109/L; platelets: <124 x 109/ L hemoglobin: <10.5 g/dL
9. Treatment with marketed or over-the-counter Vitamin D at the time of Screening (V1C) and unwilling to abstain from such medication during the 120 days when the patient will be supplemented with the trial-provided Vitamin D. A patient currently taking Vitamin D at the time of Screening (V1C) must be willing to switch to the trial-provided Vitamin D treatment and to administer it per the trial requirements.
10. (US ONLY) History of hyperparathyroidism, hypercalcemia and/or nephrolithiasis, unless appropriately treated, or any other contraindication to use of Vitamin D.
11. Any clinically significant history of an acute reaction to a vaccine or its constituents (e.g., Alhydrogel).
12. Treatment with any (live or inactive) vaccine, including influenza vaccine and Coronavirus Disease 2019 (COVID-19) vaccine, within 4 weeks prior to planned first trial dose of trial drug; or planned treatment with any vaccine up to 4 weeks after the last injection with trial drug.
13. Any acute or chronic skin infection or condition that would preclude intralymphatic injection.
14. Recent (past 12 months) or current treatment with Teplizumab (TZIELD®) or with immunosuppressant therapy, including chronic use of systemic glucocorticoid therapy. Inhaled, topical, and intranasal steroid use is acceptable. Short courses (e.g., ≤5 days) of oral, intra-articular injections or injections of steroids will be permitted during the trial.
15. Continuous/chronic treatment with prescribed or over-the-counter anti-inflammatory therapies. Short-term use (e.g., <7 days) is permissible, for example to treat a headache or in connection with a fever.
16. Known or suspected acute infection, including COVID-19 or influenza, at the time of Randomization or within 4 weeks prior to Randomization.
17. A history of epilepsy, head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles.
18. Known diagnosis of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection. Patients with previous hepatitis C infection that is now cured may be eligible.
19. Any clinically significant concomitant medical condition, including but not limited to other autoimmune diseases, cardiovascular, gastrointestinal, hematological, immune, renal including a history of renal transplantation, neurological (including Batten disease), significant diabetes complication, any underlying conditions or receiving treatments that could affect red blood cell turnover or other diseases that in the opinion of the investigator would interfere with trial participation or procedures. Celiac disease or elevated transglutaminase antibody titers is not a reason for exclusion.

    (US ONLY) Any clinically significant concomitant medical condition, including but not limited to other autoimmune or immune deficiency diseases (e.g., sarcoidosis, rheumatoid arthritis, moderate-to-severe psoriasis, inflammatory bowel disease, and other autoimmune conditions that may require treatment with TNF-alpha inhibitors or other biologics), gastrointestinal, hematological, or renal diseases including a history of any organ transplant (including renal transplantation and islet transplantation), neurological disease (including Batten disease); significant diabetes complication; a history of adrenal insufficiency; any underlying conditions or receiving treatments that could affect red blood cell turnover or other diseases that interfere with trial participation or procedures. Celiac disease or elevated transglutaminase antibody titers is not a reason for exclusion, as well as autoimmune thyroid disease under certain conditions (see Exclusion Criterion #23).
20. (US ONLY) Significant cardiovascular disease (including inadequately controlled hypertension [resting blood pressure >140/90 mmHg despite treatment], history of myocardial infarction, angina, use of anti-anginal medicines [e.g., nitroglycerin], or abnormal cardiac stress test.
21. History of significant hepatic disease or Screening alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) or aspartate aminotransferase (AST) 3 x ULN and/or total bilirubin >2 x ULN. Patients with documented Gilbert syndrome and total bilirubin level ≥2 x ULN due to unconjugated hyperbilirubinemia, without other hepatic impairment, are permitted.
22. Estimated glomerular filtration rate (eGFR) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) for those >18 years, or by the Schwartz equation for those 12 to 18 years old, <60 mL/min per 1.73 m or rapidly progressing renal disease.
23. Patients diagnosed with hypothyroidism or hyperthyroidism must be on stable treatment for at least 3 months prior to Randomization (with normal free thyroxine [T4] levels if hypothyroid).

    (US ONLY) Patients diagnosed with hypothyroidism or hyperthyroidism must be on stable treatment for at least 3 months prior to Randomization (with normal free thyroxine [T4] levels if hypothyroid). A thyroid-stimulating hormone (TSH) level > 1.5 times the ULN at Screening (V1B) is an exclusion criterion.
24. Any clinically significant abnormal findings during Screening, and any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety or ability to complete the trial.

    (US ONLY) Any clinically significant abnormal findings during Screening, and any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety or ability to complete the trial. This includes anticipated major surgery during the duration of the trial, which could interfere with participation in the trial.
25. History of malignancy not in remission within the last 5 years other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
26. Patients with any mental condition rendering him/her unable to understand the nature, scope and possible consequences of the trial, and/or evidence of poor compliance with medical instructions at Screening or showing non-compliance during the Run-In Period.
27. A history of alcohol or drug abuse or dependence within the past 12 months based on DSM IV criteria.
28. Previous treatment with the active substance recombinant human GAD65.
29. Participation in a clinical trial involving administration of an investigational drug in the past 3 months or 5 half-lives (whichever is longer) prior to first dosing of trial drug or during the trial.
30. Females who are breastfeeding, pregnant or plan to become pregnant during the trial.
31. Patients who in the opinion of the investigator will not be able to follow instructions and/or follow the trial procedures or patients that are unwilling or unable to comply with the provisions of this protocol.
32. An employee or immediate family member of an employee of Diamyd Medical AB.
33. (US ONLY)For subjects aged 18 years and older, a body mass index (BMI) ≥30 kg/m2 or ≤18.5 kg/m2; for subjects aged under 18 years BMI ≥95th percentile or ≤5th percentile for age and sex according to the US Centre for Disease Control and Prevention at V1B. (For subjects aged 18 years and older with a BMI ≥25 to ≤30 kg/m2, and for subjects aged under 18 years with a BMI ≥85th to ≤95th percentile, re-confirmation of Type 1 Diabetes diagnoses by an external, independent endocrinologist is required prior to randomization.)

Ages: 12 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Beta cell function | Baseline to 24 months
  Change from baseline to Month 24 in C-peptide area under the curve (AUC) mean 0-120 min during a 2-hour mixed meal tolerance test (MMTT)
Glycemic control | Baseline to 24 months
  Change from baseline to Month 24 in hemoglobin A1c (HbA1c).

SECONDARY OUTCOMES:
Change in time in glycemic target range 3.9 to 10 mmol/L (70 to 180 mg/dL) between baseline and Month 24. | Baseline and 24 months
  Change in time in glycemic target range 3.9 to 10 mmol/L (70 to 180 mg/dL) [evaluated from continuous glucose monitoring (CGM) data] between baseline and Month 24.
Proportion of patients with insulin dose-adjusted HbA1c ≤9 at Month 24. | 24 Months
  Proportion of patients with insulin dose-adjusted HbA1c (IDDA1C) ≤9 at Month 24.
Number of episodes per patient of severe hypoglycemia between baseline and Month 24. | Baseline and 24 months
  Number of episodes per patient of severe hypoglycemia between baseline and Month 24.
Number of episodes per patient of diabetic ketoacidosis between baseline and Month 24. | Baseline and 24 months
  Number of episodes per patient of diabetic ketoacidosis between baseline and Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, Professor, Principal Investigator — Crown Princess Victoria Children´s Hospital and Linköping University
Locations (60):
- United States (13):
  - Mary and Dick Allen Diabetes Center at Hoag Hospital, Newport Beach, California
  - Stanford University School of Medicine Center for Academic Medicine, Palo Alto, California
  - UCSD/ Rady Children's Hospital, San Diego, California
  - University of Colorado Anschutz Medical Campus, Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Diabetes Research Institute (DRI)-University of Miami Leonard M. Miller School of Medicine (UMMSM), Miami, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Washington University Diabetes Center at Barnes Jewish Hospital, St Louis, Missouri
  - Hassenfeld Children's Hospital at NYU Langone Health, Pediatric Diabetes Center, New York, New York
  - Amarillo Medical Specialists, Amarillo, Texas
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
- Czechia (4):
  - Nemocnice Jihlava, příspěvková organizace, Jihlava
  - Institut klinické a experimentální medicíny, Prague
  - Fakultní nemocnice v Motole, Prague
  - Krajská zdravotní, a.s. - Masarykova nemocnice v Ústí nad Labem, o.z., Ústí nad Labem
- Estonia (4):
  - Liina Viitas OÜ, Pärnu
  - North-Estonian Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
  - Tartu University Hospital, Children's Clinic, Tartu
- Germany (4):
  - Diabetespraxis Dr. Braun, Berlin
  - Diabetologische Schwerpunktpraxis Dres. Klaus, Dortmund
  - DZDM - Diabeteszentrum Duisburg Mitte, Duisburg
  - Justus-Liebig-Universität Gießen, Giessen
- Hungary (5):
  - Óbudai Egészségügyi Centrum, Budapest
  - Heim Pál Országos Gyermekgyógyászati Intézet, Diabetológia, Budapest
  - Észak-Budai Szent János Centrumkórház, Kútvölgyi Kórház, Belgyógyászat, Budapest
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi, Oktatókórház, Jósa András Oktatókórház, Gyermekosztály, Nyíregyháza
  - Markusovszky Egyetemi Oktatókórház, Diabetológiai Szakrendelés, Szombathely
- Netherlands (6):
  - CTU Vasculaire Geneeskunde, Locatie Academic Medical Center (AMC), Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Bethesda Diabetes Research Center te Hoogeveen, Hoogeveen
  - Dept. of Nephrology / Dept. of Endocrinology, Leiden University Medical Center (LUMC), Leiden
  - Vivendia, Nijmegen
  - Diabeter Nederland te Rotterdam, Rotterdam
- Poland (8):
  - Uniwersytecki Dziecięcy Szpital Kliniczny im. L. Zamenhofa w Białymstoku, Klinika Pediatrii, Endokrynologii, Diabetologii z Pododdziałem Kardiologii, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Klinika Pediatrii, Diabetologii i Endokrynologii, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Chorób Metabolicznych i Diabetologii, Krakow
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin
  - Kliniczny Szpital Wojewódzki nr 2 im. Św. Jadwigi Królowej w Rzeszowie, II Klinika Pediatrii, Endokrynologii i Diabetologii Dziecięcej, Rzeszów
  - Instytut Diabetologii Sp. z o.o, Warsaw
  - Panstwowy Instytut Medyczny MSWiA Klinika Chorob Wewnetrznych, Endokrynologii i Diabetologii, Warsaw
  - Instytut Pomnik - Centrum Zdrowia Dziecka (IPCZD) Oddział Diabetologii, Warsaw
- Spain (12):
  - Hospital De Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Sant Joan de Déu - Esplugues De Llobregat, Barcelona, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Complejo Hospitalario Insular de Gran Canaria, Las Palmas
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (4):
  - Skånes universitetssjukhus, Malmo, Skåne County
  - Akademiskt Specialistcentrum, Centrum for Diabetes, Stockholm, Stockholm County
  - Barn-och Ungdomscentrum Västerbotten, Norrlands Universitetssjukhus, Umeå, Västerbotten County
  - H.K.H Kronprinsessan Victorias Barn-och Ungdomssjukhus, Universitetssjukhuset i Linköping, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludvigsson J, Eriksson L, Nowak C, Teixeira PF, Widman M, Lindqvist A, Casas R, Lind M, Hannelius U. Phase III, randomised, double-blind, placebo-controlled, multicentre trial to evaluate the efficacy and safety of rhGAD65 to preserve endogenous beta cell function in adolescents and adults with recently diagnosed type 1 diabetes, carrying the genetic HLA DR3-DQ2 haplotype: the DIAGNODE-3 study protocol. BMJ Open. 2022 Oct 31;12(10):e061776. doi: 10.1136/bmjopen-2022-061776. PMID 36316084
- See also: Study website — https://diagnode-3.com/